CLINICAL TRIAL: NCT02710721
Title: Clinical Study on the Efficacy of Fasting and Nutritional Therapy as a Complementary Treatment of Advanced Metastatic Prostate Cancer Undergoing Chemotherapy - an Exploratory Randomized Controlled Trial
Brief Title: Fasting and Nutritional Therapy in Patients With Advanced Metastatic Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ProstateDiet
Record Dates: First submitted 2016-02-09; First posted 2016-03-17 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Fasting; Prostatic Neoplasms
Keywords: Fasting; Prostatic Neoplasms; Complementary Therapies; Urology
MeSH Terms: conditions — Fasting; Prostatic Neoplasms | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting (Experimental): 60h-modified fasting (36h before and 24h after chemotherapy)
  Interventions: Other: Fasting
- Control (Active Comparator): mediterranean diet
  Interventions: Other: Control

INTERVENTIONS:
Other: Fasting — Patients realize a 60h-modified fasting (36h before and 24h after chemotherapy) with a dietary energy supply 350-400kcal per day with fruit and vegetable juices or, if not feasible, an established fasting-mimicking diet of 600-800 kcal according to Longo et al. Between chemotherapy a Mediterranean diet with nutrition training individually and in small groups by trained nutritionists at the Study Centre will be practiced.
  Arms: Fasting
Other: Control — Participants of the control group will receive an individual nutrition training and in small groups according to the Mediterranean diet.
  Arms: Control

SUMMARY:
The aim of this trial is a first evaluation of the effectiveness of intermittent fasting as a supplementary therapy in patients with CRPC or hormone-sensitive prostate cancer with high metastatic load (1≥ visceral and ≥4 osseous metastases) in respect to quality of life, reduction of side effects and possible reduction in tumor progression.

DETAILED DESCRIPTION:
Prostate cancer is in Germany with approximately 25% of all cancers the most common cancer among man. Assumably there will be an increase in prostate cancer in the next few years because of demographic factors. The progressive metastatic prostate cancer often develops an androgen resistance. This so-called Castration-Resistant Prostate Cancer (CRPC) is not responsive to androgen deprivation therapy. Depending on symptoms and progression first-line chemotherapy - docetaxel and abiraterone are available.

Intermittent fasting as a form of caloric restriction has been studied most extensively experimentally in recent years. It showed consistent beneficial effects on relevant inflammatory and oncological pathways. In the field of preclinical oncology research groups have recently focused on intermittent fasting with chemotherapeutic treatment and promising experimental data have been published. In summary, the combination of fasting and chemotherapy was more effective in various cancer animal models than chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CRPC or hormone-sensitive prostate cancer with high metastatic load
* Cancer is treated to guidelines conventionally with chemotherapy or with a combination of hormone therapy and chemotherapy.

Exclusion Criteria:

* Underweight (BMI <20 kg/m2) or actual weight decrease >2 kg or >5 kg in the last 1 or 3 months.
* Eating disorder
* Dementia
* Psychosis
* Terminal illness with a significant limitation of mobility and overall vitality
* Diabetes mellitus type 1
* Renal insufficiency stage > 2, GFR <60mlmin / 1.73 m2

Ages: 25 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
FACT-P/-Taxane/-An sum score | Assessment day 0 (baseline) and 7 days after each of 6 chemotherapies (study weeks 1,4,7,10,13,16)
  summarized change of FACT score from baseline to day 8 after each chemotherapy

SECONDARY OUTCOMES:
FACT-P/-Taxane/-An sum score | Assessment day 0 (baseline) and 3 and 6 months after day 0
  Change of score after 3 and 6 months
HADS | Assessment day 0 (baseline) and 7 days after each of 6 chemotherapies (study weeks 1,4,7,10,13,16) and after 3 and 6 months after study day 0
  Summarized change of score for all time Points

OTHER OUTCOMES:
Differential blood count | Assessment day 0 (baseline) and 7 days after each of 6 chemotherapies (study weeks 1,4,7,10,13,16) and after 3 and 6 months after study day 0
  Summarized changes of blood count
Intensity of chemotherapy- related side effects | Assessment day 0 (baseline) and 7 days after each of 6 chemotherapies (study weeks 1,4,7,10,13,16)
  Group difference of summarized frequency and intensity

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite Centrum Epidemiologie und Gesundheitsökonomie, CC1: Gesundheitswissenschaften; Kurt Miller, Prof. Dr., Principal Investigator — Charité Centrum Chirurgische Medizin, CC 8 Klinik für Urologie; Ursula Steiner, Dr., Principal Investigator — Charité Centrum Chirurgische Medizin, CC 8 Klinik für Urologie
Locations (1):
- Charité Centrum Chirurgische Medizin, CC 8 Klinik für Urologie, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided